CLINICAL TRIAL: NCT02824198
Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine Given as a Booster Injection in Adolescents and Adults Who Previously Completed the 3-dose Schedule in a Study Conducted in Singapore
Brief Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine Booster Injection in Subjects Who Previously Completed a 3-dose Schedule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CYD63; U1111-1161-2813 (Other: WHO)
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Hemorrhagic Fever; Dengue Virus; CYD Dengue Vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Dosage Forms; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: An observer-blind procedure was followed for the injection of CYD dengue vaccine or placebo. Neither the blind-observer Investigator nor the participants (and/or participants' parent(s)/legally acceptable representative(s) for participants aged < 21 years) knew which product was administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYD Dengue Vaccine booster Group (Experimental): Participants who received 3 doses of the tetravalent dengue vaccine in a previous CYD dengue vaccine study (CYD28), received a booster injection of CYD dengue vaccine at Day 0 in this study (CYD63).
  Interventions: Biological: CYD Dengue Vaccine (5 dose formulation)
- Placebo Group (Placebo Comparator): Participants who received 3 doses of the tetravalent dengue vaccine in a previous CYD dengue vaccine study (CYD28), received an injection of a placebo at Day 0 in this study (CYD63).
  Interventions: Biological: Placebo, NaCl 0.9%

INTERVENTIONS:
Biological: CYD Dengue Vaccine (5 dose formulation) — 0.5 mL, Subcutaneous
  Arms: CYD Dengue Vaccine booster Group
Biological: Placebo, NaCl 0.9% — 0.5 mL, Subcutaneous
  Arms: Placebo Group

SUMMARY:
The aim of the study was to assess and describe the booster effect of a tetravalent CYD dengue vaccine dose administered about 5 years or more after the completion of a 3-dose vaccination schedule in Singapore.

Primary Objective:

* To demonstrate the non-inferiority in terms of geometric mean of titer ratios (GMTRs) of a CYD dengue vaccine booster compared to the third CYD dengue vaccine injection in participants from CYD28 trial (participants from Group 1 only).

Secondary Objectives:

* If the primary objective of non-inferiority achieved: To demonstrate the superiority, in terms of GMTRs, of a CYD dengue vaccine booster compared to the third CYD dengue vaccine injection in participants from CYD28 trial (participants from Group 1 only).
* To describe the immune responses elicited by the CYD dengue vaccine booster or placebo injection in participants who received three doses of the CYD dengue vaccine in the CYD28 trial in all participants.
* To describe the neutralizing antibody levels of each dengue serotype Post Dose 3 (CYD28 participants) and immediately prior to booster or placebo injection in all participants.
* To describe the neutralizing antibody persistence 6 months, 1 year and 2 years post booster or placebo injection in all study participants.
* To evaluate the safety of booster vaccination with CYD dengue vaccine in all participants.

DETAILED DESCRIPTION:
Healthy adolescents and adults received 3 doses of the tetravalent dengue vaccine 5-6 years earlier in a previous CYD dengue vaccine trial (CYD28 - NCT00880893) received either a booster injection of CYD dengue vaccine or a placebo on Day 0. They were evaluated for safety and antibody persistence of the booster injection up to 2 years post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Had been identified as a potential participant by the Sponsor, and was included in the list provided to the investigator (i.e., aged 9 to 45 years on the day of first injection of CYD dengue vaccine in CYD28, had received 3 doses of CYD dengue vaccine in the CYD28 trial, and had a post-dose 3 serum sample available).
* Participants with good health, based on medical history and physical examination.
* Informed consent form (ICF) had been signed and dated by participant (based on local regulations), and ICF had been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations).
* Participant and parent(s)/legally acceptable representative(s) was able to attend all scheduled visits to comply with all trial procedures.

Exclusion Criteria:

* Participant who received any other dengue vaccination that was not part of CYD28.
* Participant was pregnant, or lactating, or of childbearing potential (considered of non childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination).
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following the trial vaccination
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0°C). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-03-18 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Park J, Archuleta S, Oh MH, Shek LP, Jin J, Bonaparte M, Fargo C, Bouckenooghe A. Immunogenicity and safety of a dengue vaccine given as a booster in Singapore: a randomized Phase II, placebo-controlled trial evaluating its effects 5-6 years after completion of the primary series. Hum Vaccin Immunother. 2020 Mar 3;16(3):523-529. doi: 10.1080/21645515.2019.1661204. Epub 2019 Nov 5. PMID 31464558
- [Derived] Park J, Archuleta S, Oh MH, Shek LP, Wang H, Bonaparte M, Frago C, Bouckenooghe A, Jantet-Blaudez F, Begue S, Gimenez-Fourage S, Pagnon A. Humoral and cellular immunogenicity and safety following a booster dose of a tetravalent dengue vaccine 5+ years after completion of the primary series in Singapore: 2-year follow-up of a randomized phase II, placebo-controlled trial. Hum Vaccin Immunother. 2021 Jul 3;17(7):2107-2116. doi: 10.1080/21645515.2020.1861875. Epub 2021 Feb 24. PMID 33626291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 01 July 2016 to 18 February 2017 at 3 sites in Singapore.
Pre-assignment Details: A total of 118 participants who received 3 doses of CYD dengue vaccine in study CYD28 (NCT00880893) were enrolled and randomized in this study (CYD63).
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Started | 89 | 29
Completed | 74 | 26
Not Completed | 15 | 3
Not completed — Non-compliance with the protocol | 5 | 1
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group | Total
Number analyzed (Participants) | 89 | 29 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 0 | 11
  Between 18 and 65 years | 78 | 29 | 107
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (11.18) | 28.2 (9.18) | 28.2 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 15 | 58
  Male | 46 | 14 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Each Dengue Virus Serotype Following Booster Injection With CYD Dengue Vaccine in CYD63 Compared to the Third CYD Dengue Vaccine Injection Received in Study CYD28: CYD Dengue Vaccine Booster Group
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) were assessed using the plaque reduction neutralization test (PRNT).
Time Frame: 28 days post-dose 3 in CYD28 and 28 days post-booster injection in CYD63
Population: Analysis was performed on Per-Protocol Analysis Set which included all participants who had no protocol deviations from the present study (CYD63). Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- CYD Dengue Vaccine Booster Group: Post Dose 3 in CYD28: Participants who received 3 doses of tetravalent dengue vaccine in previous study (CYD28) were enrolled in this study (CYD63).
- CYD Dengue Vaccine Booster Group: Post Booster Dose: Participants who received 3 doses of the tetravalent dengue vaccine in a previous CYD dengue vaccine study (CYD28), received a booster injection of CYD dengue vaccine at Day 0 in this study (CYD63).
Arm/Group | CYD Dengue Vaccine Booster Group: Post Dose 3 in CYD28 | CYD Dengue Vaccine Booster Group: Post Booster Dose
Number analyzed (Participants) | 75 | 75
titers (1/dilution)
  Dengue Virus Serotype 1: number analyzed (Participants) | 74 | 75
  Dengue Virus Serotype 1 | 20.3 [13.9 to 29.5] | 37.7 [26.4 to 53.7]
  Dengue Virus Serotype 2: number analyzed (Participants) | 73 | 75
  Dengue Virus Serotype 2 | 85.6 [55.7 to 132] | 56.2 [38.5 to 82.1]
  Dengue Virus Serotype 3: number analyzed (Participants) | 72 | 75
  Dengue Virus Serotype 3 | 102 [78.4 to 133] | 105 [77.4 to 142]
  Dengue Virus Serotype 4: number analyzed (Participants) | 70 | 75
  Dengue Virus Serotype 4 | 92.8 [72.5 to 119] | 123 [93.8 to 161]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Booster Group: Post Dose 3 in CYD28 vs CYD Dengue Vaccine Booster Group: Post Booster Dose; Dengue Virus Serotype 1; Test type: Non-Inferiority — The overall non-inferiority of the booster dose was to be demonstrated if the lower limit of the two-sided 95% Confidence Interval (CI) of the Geometric mean of titer ratios (GMTRs) (booster vs post-dose 3) was greater than (>) 1/2 for each serotype; Geometric mean of titer ratio = 1.34, 95% CI 2-sided [0.998 to 1.79]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Booster Group: Post Dose 3 in CYD28 vs CYD Dengue Vaccine Booster Group: Post Booster Dose; Dengue Virus Serotype 2; Test type: Non-Inferiority — The overall non-inferiority of the booster dose was to be demonstrated if the lower limit of the two-sided 95% CI of the GMTRs (booster vs post-dose 3) was > 1/2 for each serotype; Geometric mean of titer ratio = 0.603, 95% CI 2-sided [0.439 to 0.829]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Booster Group: Post Dose 3 in CYD28 vs CYD Dengue Vaccine Booster Group: Post Booster Dose; Dengue Virus Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Geometric mean of titer ratio = 0.979, 95% CI 2-sided [0.746 to 1.28]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Booster Group: Post Dose 3 in CYD28 vs CYD Dengue Vaccine Booster Group: Post Booster Dose; Dengue Virus Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Geometric mean of titer ratio = 1.27, 95% CI 2-sided [0.918 to 1.75]

2. Secondary Outcome: GMTs of Antibodies Against Each Dengue Virus Serotype Before and Following Booster Injection (Inj.) With Either CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) following booster injection were assessed using PRNT.
Time Frame: Pre-booster injection (Day 0) and 28 days post-booster injection
Population: Analysis was performed on Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
titers (1/dilution)
  Dengue Virus Serotype 1: Pre-booster Inj. | 13.5 [9.31 to 19.6] | 16.7 [7.73 to 36.1]
  Dengue Virus Serotype 1: 28 days Post-booster Inj. | 37.7 [26.4 to 53.7] | 18.1 [8.61 to 38.1]
  Dengue Virus Serotype 2: Pre-booster Inj. | 18.4 [12.1 to 28.0] | 23.2 [9.97 to 53.9]
  Dengue Virus Serotype 2: 28 days Post-booster Inj. | 56.2 [38.5 to 82.1] | 21.5 [9.61 to 48.1]
  Dengue Virus Serotype 3: Pre-booster Inj. | 22.4 [15.6 to 32.0] | 27.4 [14.8 to 51.0]
  Dengue Virus Serotype 3: 28 days Post-booster Inj. | 105 [77.4 to 142] | 24.1 [13.6 to 42.6]
  Dengue Virus Serotype 4: Pre-booster Inj. | 28.0 [20.4 to 38.5] | 44.9 [28.3 to 71.3]
  Dengue Virus Serotype 4: 28 days Post-booster Inj. | 123 [93.8 to 161] | 39.8 [23.9 to 66.3]

3. Secondary Outcome: GMTRs of Antibodies Against Each Dengue Virus Serotype Before and Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) following booster injection were assessed using PRNT. GMTRs were calculated as the ratio of GMTs post-booster injection and pre-booster injection.
Time Frame: Pre-booster injection (Day 0) and 28 days post-booster injection
Population: Analysis was performed on Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
ratio
  Dengue Virus Serotype 1 | 1.74 [1.33 to 2.28] | 0.676 [0.525 to 0.871]
  Dengue Virus Serotype 2 | 2.04 [1.54 to 2.69] | 0.624 [0.523 to 0.745]
  Dengue Virus Serotype 3 | 3.52 [2.58 to 4.82] | 0.669 [0.513 to 0.873]
  Dengue Virus Serotype 4 | 3.58 [2.61 to 4.90] | 0.822 [0.640 to 1.06]

4. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Before and Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Seropositivity against each dengue virus serotype were measured using dengue PRNT. Seropositive participants were defined as the participants with neutralizing antibody titers >=10 (1/dilution).
Time Frame: Pre-booster injection (Day 0) and 28 days post-booster injection
Population: Analysis was performed on Per-Protocol Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
percentage of participants
  Dengue Virus Serotype 1: Pre-booster Inj. | 32.0 | 32.1
  Dengue Virus Serotype 1: 28 days Post-booster Inj. | 74.7 | 35.7
  Dengue Virus Serotype 2: Pre-booster Inj. | 41.3 | 42.9
  Dengue Virus Serotype 2: 28 days Post-booster Inj. | 81.3 | 42.9
  Dengue Virus Serotype 3: Pre-booster Inj. | 58.7 | 60.7
  Dengue Virus Serotype 3: 28 days Post-booster Inj. | 96.0 | 67.9
  Dengue Virus Serotype 4: Pre-booster Inj. | 70.7 | 89.3
  Dengue Virus Serotype 4: 28 days Post-booster Inj. | 97.3 | 82.1

5. Secondary Outcome: Percentage of Participants With Seroconversion Against Each Dengue Virus Serotype Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Seroconversion rates for each serotypes were defined as the percentages of participants with either a pre-booster titer < 10 (1/dilution) and a post-booster titer >= 40 (1/dilution), or a pre-booster titer >=10 (1/dilution) and a >= 4-fold increase in post-booster titer as determined by PRNT.
Time Frame: 28 days post-booster injection
Population: Analysis was performed on Per-Protocol Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
percentage of participants
  Dengue Virus Serotype 1 | 29.3 | 3.6
  Dengue Virus Serotype 2 | 29.3 | 0.0
  Dengue Virus Serotype 3 | 44.0 | 0.0
  Dengue Virus Serotype 4 | 38.7 | 0.0

6. Secondary Outcome: GMTs of Antibodies Against Each Dengue Virus Serotype Following the Third CYD Dengue Vaccine Injection Received In Study CYD28 and Before Booster Injection With Either CYD Dengue Vaccine or Placebo in CYD63
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) were assessed using the PRNT.
Time Frame: 28 days post-dose 3 in CYD28 and pre-booster injection (Day 0) in CYD 63
Population: Analysis was performed on Per-Protocol Analysis Set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
titers (1/dilution)
  Dengue Virus Serotype 1: 28 days Post-dose 3: number analyzed (Participants) | 74 | 28
  Dengue Virus Serotype 1: 28 days Post-dose 3 | 20.3 [13.9 to 29.5] | 26.8 [12.4 to 57.7]
  Dengue Virus Serotype 1: Pre-booster Inj. | 13.5 [9.31 to 19.6] | 16.7 [7.73 to 36.1]
  Dengue Virus Serotype 2: 28 days Post-dose 3: number analyzed (Participants) | 73 | 27
  Dengue Virus Serotype 2: 28 days Post-dose 3 | 85.6 [55.7 to 132] | 65.4 [28.3 to 151]
  Dengue Virus Serotype 2: Pre-booster Inj. | 18.4 [12.1 to 28.0] | 23.2 [9.97 to 53.9]
  Dengue Virus Serotype 3: 28 days Post-dose 3: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 3: 28 days Post-dose 3 | 102 [78.4 to 133] | 107 [63.6 to 179]
  Dengue Virus Serotype 3: Pre-booster Inj. | 22.4 [15.6 to 32.0] | 27.4 [14.8 to 51.0]
  Dengue Virus Serotype 4: 28 days Post-dose 3: number analyzed (Participants) | 70 | 26
  Dengue Virus Serotype 4: 28 days Post-dose 3 | 92.8 [72.5 to 119] | 86.5 [51.0 to 147]
  Dengue Virus Serotype 4: Pre-booster Inj. | 28.0 [20.4 to 38.5] | 44.9 [28.3 to 71.3]

7. Secondary Outcome: GMTRs of Antibodies Against Each Dengue Virus Serotype Following the Third CYD Dengue Vaccine Injection Received in Study CYD28 And Before Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) were assessed using the PRNT. GMTRs were calculated as the ratio of GMTs post-dose 3 in CYD28 and pre-booster injection in CYD63.
Time Frame: 28 days post-dose 3 in CYD28 and pre-booster injection (Day 0) in CYD63
Population: Analysis was performed on Per-Protocol Analysis Set. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
ratio
  Dengue Virus Serotype 1: number analyzed (Participants) | 74 | 28
  Dengue Virus Serotype 1 | 0.487 [0.390 to 0.609] | 0.441 [0.316 to 0.617]
  Dengue Virus Serotype 2: number analyzed (Participants) | 73 | 27
  Dengue Virus Serotype 2 | 0.199 [0.160 to 0.248] | 0.313 [0.224 to 0.437]
  Dengue Virus Serotype 3: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 3 | 0.207 [0.163 to 0.262] | 0.267 [0.171 to 0.416]
  Dengue Virus Serotype 4: number analyzed (Participants) | 70 | 26
  Dengue Virus Serotype 4 | 0.291 [0.217 to 0.391] | 0.474 [0.343 to 0.656]

8. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Following the Third CYD Dengue Vaccine Injection Received in Study CYD28, and Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: as for outcome 4
Time Frame: 28 days post-dose 3 in CYD28 and 28 days post-booster injection in CYD63
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
percentage of participants
  Dengue Virus Serotype 1: 28 days Post-dose 3: number analyzed (Participants) | 74 | 28
  Dengue Virus Serotype 1: 28 days Post-dose 3 | 52.7 | 50.0
  Dengue Virus Serotype 1: 28 days Post-booster Inj. | 74.7 | 35.7
  Dengue Virus Serotype 2: 28 days Post-dose 3: number analyzed (Participants) | 73 | 27
  Dengue Virus Serotype 2: 28 days Post-dose 3 | 89.0 | 74.1
  Dengue Virus Serotype 2: 28 days Post-booster Inj. | 81.3 | 42.9
  Dengue Virus Serotype 3: 28 days Post-dose 3: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 3: 28 days Post-dose 3 | 97.2 | 96.3
  Dengue Virus Serotype 3: 28 days Post-booster Inj. | 96.0 | 67.9
  Dengue Virus Serotype 4: 28 days Post-dose 3: number analyzed (Participants) | 70 | 26
  Dengue Virus Serotype 4: 28 days Post-dose 3 | 95.7 | 88.5
  Dengue Virus Serotype 4: 28 days Post-booster Inj. | 97.3 | 82.1

9. Secondary Outcome: GMTs of Antibodies Against Each Dengue Virus Serotype Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: as for outcome 2
Time Frame: 6 months, 12 months, and 24 months post-booster injection
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
titers (1/dilution)
  Dengue Virus Serotype 1:6 months Post-booster Inj.: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 1:6 months Post-booster Inj. | 25.1 [17.4 to 36.4] | 14.3 [7.42 to 27.6]
  Dengue Virus Serotype1:12 months Post-booster Inj.: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype1:12 months Post-booster Inj. | 20.9 [14.0 to 31.1] | 14.6 [7.55 to 28.3]
  Dengue Virus Serotype1:24 months Post-booster Inj.: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype1:24 months Post-booster Inj. | 14.4 [9.88 to 21.0] | 13.6 [7.14 to 25.7]
  Dengue Virus Serotype 2:6 months Post-booster Inj.: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 2:6 months Post-booster Inj. | 44.3 [29.0 to 67.7] | 20.4 [9.07 to 45.9]
  Dengue Virus Serotype2:12 months Post-booster Inj.: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype2:12 months Post-booster Inj. | 39.3 [25.3 to 61.2] | 22.1 [9.95 to 49.1]
  Dengue Virus Serotype2:24 months Post-booster Inj.: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype2:24 months Post-booster Inj. | 41.6 [25.8 to 67.2] | 21.7 [9.49 to 49.8]
  Dengue Virus Serotype 3:6 months Post-booster Inj.: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 3:6 months Post-booster Inj. | 65.1 [47.3 to 89.5] | 26.7 [15.3 to 46.7]
  Dengue Virus Serotype3:12 months Post-booster Inj.: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype3:12 months Post-booster Inj. | 54.8 [40.1 to 74.9] | 20.6 [11.8 to 36.0]
  Dengue Virus Serotype3:24 months Post-booster Inj.: number analyzed (Participants) | 65 | 26
  Dengue Virus Serotype3:24 months Post-booster Inj. | 36.5 [25.6 to 51.8] | 16.8 [9.36 to 30.2]
  Dengue Virus Serotype 4:6 months Post-booster Inj.: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 4:6 months Post-booster Inj. | 75.6 [58.8 to 97.2] | 34.6 [20.5 to 58.5]
  Dengue Virus Serotype4:12 months Post-booster Inj.: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype4:12 months Post-booster Inj. | 61.9 [47.2 to 81.2] | 33.1 [21.0 to 52.2]
  Dengue Virus Serotype4:24 months Post-booster Inj.: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype4:24 months Post-booster Inj. | 50.1 [38.4 to 65.4] | 24.5 [14.0 to 42.8]

10. Secondary Outcome: GMTRs of Antibodies Against Each Dengue Virus Serotype Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: as for outcome 3
Time Frame: Pre-booster injection (Day 0) and 6 months, 12 months, 24 months post-booster injection
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
ratio
  Dengue Virus Serotype 1: 6 months/Day 0: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 1: 6 months/Day 0 | 1.19 [0.953 to 1.51] | 0.646 [0.544 to 0.767]
  Dengue Virus Serotype 1: 12 months/Day 0: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype 1: 12 months/Day 0 | 0.983 [0.775 to 1.25] | 0.660 [0.516 to 0.845]
  Dengue Virus Serotype 1: 24 months/Day 0: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype 1: 24 months/Day 0 | 0.658 [0.528 to 0.818] | 0.594 [0.500 to 0.705]
  Dengue Virus Serotype 2: 6 months/Day 0: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 2: 6 months/Day 0 | 1.60 [1.25 to 2.06] | 0.634 [0.525 to 0.766]
  Dengue Virus Serotype 2: 12 months/Day 0: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype 2: 12 months/Day 0 | 1.42 [1.11 to 1.80] | 0.687 [0.564 to 0.838]
  Dengue Virus Serotype 2: 24 months/Day 0: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype 2: 24 months/Day 0 | 1.43 [1.12 to 1.84] | 0.646 [0.491 to 0.850]
  Dengue Virus Serotype 3: 6 months/Day 0: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 3: 6 months/Day 0 | 2.14 [1.60 to 2.85] | 0.797 [0.606 to 1.05]
  Dengue Virus Serotype 3: 12 months/Day 0: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype 3: 12 months/Day 0 | 1.76 [1.35 to 2.30] | 0.614 [0.455 to 0.829]
  Dengue Virus Serotype 3: 24 months/Day 0: number analyzed (Participants) | 65 | 26
  Dengue Virus Serotype 3: 24 months/Day 0 | 1.11 [0.876 to 1.42] | 0.479 [0.357 to 0.642]
  Dengue Virus Serotype 4: 6 months/Day 0: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 4: 6 months/Day 0 | 2.17 [1.67 to 2.82] | 0.743 [0.530 to 1.04]
  Dengue Virus Serotype 4: 12 months/Day 0: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype 4: 12 months/Day 0 | 1.70 [1.28 to 2.27] | 0.710 [0.556 to 0.906]
  Dengue Virus Serotype 4: 24 months/Day 0: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype 4: 24 months/Day 0 | 1.35 [1.04 to 1.75] | 0.529 [0.384 to 0.730]

11. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: as for outcome 4
Time Frame: 6 months, 12 months, and 24 months post-booster injection
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 75 | 28
percentage of participants
  Dengue Virus Serotype 1:6 months Post-booster Inj.: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 1:6 months Post-booster Inj. | 59.7 | 33.3
  Dengue Virus Serotype1:12 months Post-booster Inj.: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype1:12 months Post-booster Inj. | 49.3 | 33.3
  Dengue Virus Serotype1:24 months Post-booster Inj.: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype1:24 months Post-booster Inj. | 37.9 | 34.6
  Dengue Virus Serotype 2:6 months Post-booster Inj.: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 2:6 months Post-booster Inj. | 72.2 | 40.7
  Dengue Virus Serotype2:12 months Post-booster Inj.: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype2:12 months Post-booster Inj. | 66.7 | 44.4
  Dengue Virus Serotype2:24 months Post-booster Inj.: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype2:24 months Post-booster Inj. | 65.2 | 42.3
  Dengue Virus Serotype 3:6 months Post-booster Inj.: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 3:6 months Post-booster Inj. | 88.9 | 70.4
  Dengue Virus Serotype3:12 months Post-booster Inj.: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype3:12 months Post-booster Inj. | 89.9 | 63.0
  Dengue Virus Serotype3:24 months Post-booster Inj.: number analyzed (Participants) | 65 | 26
  Dengue Virus Serotype3:24 months Post-booster Inj. | 76.9 | 50.0
  Dengue Virus Serotype 4:6 months Post-booster Inj.: number analyzed (Participants) | 72 | 27
  Dengue Virus Serotype 4:6 months Post-booster Inj. | 95.8 | 77.8
  Dengue Virus Serotype4:12 months Post-booster Inj.: number analyzed (Participants) | 69 | 27
  Dengue Virus Serotype4:12 months Post-booster Inj. | 91.3 | 85.2
  Dengue Virus Serotype4:24 months Post-booster Inj.: number analyzed (Participants) | 66 | 26
  Dengue Virus Serotype4:24 months Post-booster Inj. | 89.4 | 65.4

12. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions (Pain, Erythema, Swelling) Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Grade 3 injection site reactions: Pain: significant; prevents daily activity; Erythema and Swelling: >100 millimeter.
Time Frame: Within 7 days after booster injection
Population: Analysis was performed on Safety Analysis Set which included all participants who received either CYD dengue vaccine or placebo. Here, 'number analyzed' = participants with available data for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 89 | 29
Participants
  Injection-site Pain: Any: number analyzed (Participants) | 88 | 28
  Injection-site Pain: Any | 29 | 7
  Injection-site Pain: Grade 3: number analyzed (Participants) | 88 | 28
  Injection-site Pain: Grade 3 | 1 | 0
  Injection-site Erythema: Any: number analyzed (Participants) | 88 | 28
  Injection-site Erythema: Any | 1 | 0
  Injection-site Erythema: Grade 3: number analyzed (Participants) | 88 | 28
  Injection-site Erythema: Grade 3 | 0 | 0
  Injection-site Swelling: Any: number analyzed (Participants) | 88 | 28
  Injection-site Swelling: Any | 0 | 0
  Injection-site Swelling: Grade 3: number analyzed (Participants) | 88 | 28
  Injection-site Swelling: Grade 3 | 0 | 0

13. Secondary Outcome: Number of Participants Reporting Solicited Systemic Reactions (Fever, Headache, Malaise, Myalgia, Asthenia) Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Grade 3 reactions: Fever: >=39 degree Celsius; Headache, Malaise, Myalgia, and Asthenia: significant, prevents daily activity.
Time Frame: Within 14 days after booster injection
Population: Analysis was performed on Safety Analysis Set. Here, 'number analyzed' = participants with available data for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 89 | 29
Participants
  Fever: Any Grade: number analyzed (Participants) | 88 | 28
  Fever: Any Grade | 2 | 0
  Fever: Grade 3: number analyzed (Participants) | 88 | 28
  Fever: Grade 3 | 0 | 0
  Headache: Any Grade: number analyzed (Participants) | 88 | 28
  Headache: Any Grade | 23 | 3
  Headache: Grade 3: number analyzed (Participants) | 88 | 28
  Headache: Grade 3 | 0 | 0
  Malaise: Any Grade: number analyzed (Participants) | 88 | 28
  Malaise: Any Grade | 11 | 3
  Malaise: Grade 3: number analyzed (Participants) | 88 | 28
  Malaise: Grade 3 | 0 | 1
  Myalgia: Any Grade: number analyzed (Participants) | 88 | 28
  Myalgia: Any Grade | 21 | 7
  Myalgia: Grade 3: number analyzed (Participants) | 88 | 28
  Myalgia: Grade 3 | 0 | 1
  Asthenia: Any Grade: number analyzed (Participants) | 88 | 28
  Asthenia: Any Grade | 15 | 4
  Asthenia: Grade 3: number analyzed (Participants) | 88 | 28
  Asthenia: Grade 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected from Day 0 (post-vaccination) up to 28 days post-booster injection. Solicited Reaction (SR) data were collected within 7 and 14 days after vaccination. Serious adverse event (SAE) data were collected throughout the study (up to 24 months after booster injection).
Description: Analysis was performed on Safety Analysis Set. A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/29
Serious Adverse Events (participants affected / at risk) | 5/89 | 0/29
Other Adverse Events (participants affected / at risk) | 47/89 | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Booster Group (N=89) | Placebo Group (N=29)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Booster Group (N=89) | Placebo Group (N=29)
Asthenia (General disorders) | 15 (15) | 4 (4)
Injection Site Pain (General disorders) | 29 (29) | 7 (7)
Malaise (General disorders) | 11 (11) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (7) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (21) | 7 (7)
Headache (Nervous system disorders) | 23 (23) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT02824198/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT02824198/SAP_001.pdf